CLINICAL TRIAL: NCT04875117
Title: Investigating the Impact of Hearing Aid Fitting on Fatigue.
Brief Title: Fatigue and Hearing Loss.
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 17082
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Hearing Loss; Fatigue
MeSH Terms: conditions — Hearing Loss; Fatigue | interventions — Hearing Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Participants who are due to receive their first-ever hearing aid(s) as part of their routine audiological care.
  Interventions: Device: Hearing aid
- Control: Participants with hearing loss who have not experienced any change in hearing aid status for at least 1 year.

INTERVENTIONS:
Device: Hearing aid — One or two behind the ear hearing aids provided by the UK National Health Service.
  Groups: Intervention

SUMMARY:
An intervention group and a control group will complete a battery of questionnaires at four time points to investigate the impact of first-ever hearing aid fitting on fatigue and associated variables. The study is observational as all participants in the intervention group will already be receiving their first-ever hearing aid as part of their routine audiological care.

DETAILED DESCRIPTION:
Hearing Impairment leads to increased listening effort which could result in short and/or long term fatigue. Previous research has shown that people with a hearing loss score higher on fatigue questionnaires than people without a hearing loss. Hearing Aid fitting has been shown to reduce fatigue in an objective measurement study, however no reduction has been shown using subjective measurement. To examine the effect of hearing aid fitting on fatigue a longitudinal study will be conducted. A battery of questionnaires measuring fatigue, listening effort, daily activity, need for cognition and hearing handicap as well as an objective hearing test will be conducted at 4 time points. These time points will be a baseline assessment before hearing aid fitting, 2 weeks after fitting (~3 months after baseline), 3 months after fitting and 6 months after fitting. A control group with no change in hearing aid status will also be measured at these time points. The study is observational as all participants in the intervention group will already be receiving their first-ever hearing aid as part of their routine audiological care. This study monitors the effect of the hearing aid fitting.

The general hypothesis is that hearing aid fitting will reduce fatigue. More specifically it is expected that fatigue will increase immediately after fitting and then decrease by the 6 month time point. It is also expected that social activity levels will increase after fitting and that individual differences in this activity change will explain some of the differences between participants in rate of change in fatigue. It is predicted that high Need for Cognition and Hearing Handicap scores will increase the amount of change in fatigue for the intervention group. 57 participants will be recruited for each group, each participant being involved in the study for no more than 7 months with the study running for a total of 15 months. The data will be analysed using multi-level analysis.

ELIGIBILITY:
Inclusion Criteria:

* A self-reported hearing loss.
* Aged between 18 and 75 years old.

Inclusion criteria for intervention group only:

* Must already have an appointment arranged to receive a hearing aid for the first time.

Inclusion criteria for control group only:

* No change in hearing aid status (including new models) for the past 1 year.

Exclusion Criteria:

* Non fluent English speakers. (To maintain validity of results as English language questionnaires are used)
* Inability to read (In order to complete the questionnaires).
* Inability to visit on multiple occasions over 7 months (e.g. can't be planning to move away from the area).
* Inability to give full informed consent.
* Primary complaint of tinnitus.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population are adults with hearing loss. The intervention group are those already due to receive their first-ever hearing aid as part of their routine audiological care, while the controls experience no change in hearing aid status for at least one year.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue Assessment Scale (FAS) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of general fatigue.

SECONDARY OUTCOMES:
Change in the Multidimensional Fatigue Symptom Inventory - short form (MFSI-SF) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of general fatigue.
Change in Vanderbilt Fatigue Scale (VFS) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of listening-related fatigue.
Change in Listening Effort Assessment Questionnaire (LEAS) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of listening effort
Change in International Physical Activity Questionnaire short form (IPAQ) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of physical activity
Craig Handicap Assessment and Reporting Technique (CHART) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of work activity
Change in Social Participation Restrictions Questionnaire (SPaRQ) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of social participation restrictions
Change in Social Participation Questionnaire (SPQ) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of social activity
Change in Social activity log (SAL) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of social activity
Change in Auditory Lifestyle Demand Questionnaire (ALDQ) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of auditory lifestyle
Need for Cognition Scale (NFCS) | Once at baseline assessment only
  A self-report measure of participants' enjoyment of cognitive challenges.
Change in Hearing Handicap Inventory for Adults (HHIA) | Baseline, 3 months after baseline, 6 months after baseline and 9 months after baseline.
  A self-report measure of hearing handicap

CONTACTS AND LOCATIONS:
Overall Officials: Graham Naylor, Principal Investigator — Director
Locations (2):
- United Kingdom (2):
  - NHS audiology department, Glasgow Royal Infirmary, Glasgow
  - University of Nottingham Hearing Sciences - Scottish Section, Glasgow

IPD SHARING:
Plan to Share IPD: Undecided
All anonymised raw data are to be made available upon request.